CLINICAL TRIAL: NCT01510314
Title: Comparison of C-reactive Protein and Procalcitonin to Detect Infectious Complications After Elective Colorectal Surgery
Brief Title: Inflammatory Markers After COloRectal Surgery)
Acronym: IMACORS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: ORTEGA GGEST 2011
Record Dates: First submitted 2012-01-13; First posted 2012-01-16 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Infectious Complications After Colorectal Surgery
MeSH Terms: interventions — C-Reactive Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: C-reactive protein and procalcitonin dosages

SUMMARY:
The clinical symptoms of septic complications (SC) (responsible for the majority of morbidity in colorectal surgery) become apparent only 5-7 days after the operation, whereas the efficacy of treatment depends on early diagnosis. By detecting such complications early it could be possible to reduce their severity, the length of hospitalisation, repeat colostomy and the number of readmissions. Our team has shown that C-reactive protein (CRP) > 125 mg/L at postoperative day 4 (D4) was a predictor of SC in this context. Procalcitonin (PCT) is a marker of sepsis currently used in intensive care, but its use in the follow-up of elective surgery, particularly colorectal surgery, has not been fully evaluated.

The aim of this study is to compare the ability of CRP and PCT to detect SC as early as postoperative day 2 (D2) (intra-abdominal or systemic SC, such as those defined by the CDC) after elective colorectal surgery.

Adult patients about to undergo elective colorectal surgery with anastomosis will be included once they have given their written informed consent. Levels of CRP and PCT will be measured the day before the surgery, then at D1, D2, D3 and D4. The clinical data (temperature, recovery of bowel movement, pain, pain on palpation) will be recorded daily. Imaging examinations will be performed at the discretion of the surgeon; the only obligation will be to perform a contrast-enhanced abdominopelvic CT-scan if CRP at D4 > 125 mg/L with no other clinical anomalies. The discriminating ability (measured by the area under the ROC curve) of CRP at D2 was 0.653 in our previous study. An improvement of at least 0.1 will be necessary to show the superiority of PCT over CRP in clinical terms and with regard to the cost.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective colorectal surgery with anastomosis for benign or malignant disease
* > 18 years old
* Giving written informed consent
* Included in the national health insurance

Exclusion Criteria:

* Emergent surgery
* Previous infection
* Patients undergoing Hyperthermic Intraperitoneal Chemotherapy
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 552 (Actual)
Dates: Start 2011-11 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Intraabdominal infection

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Ortega-Deballon, Principal Investigator — Centre Hospitalier Universitaire Dijon
Locations (3):
- France (3):
  - CHU Besançon, Besançon
  - CGFL, Dijon
  - CHU Dijon, Dijon

REFERENCES:
- [Result] Facy O, Paquette B, Orry D, Binquet C, Masson D, Bouvier A, Fournel I, Charles PE, Rat P, Ortega-Deballon P; IMACORS Study. Diagnostic Accuracy of Inflammatory Markers As Early Predictors of Infection After Elective Colorectal Surgery: Results From the IMACORS Study. Ann Surg. 2016 May;263(5):961-6. doi: 10.1097/SLA.0000000000001303. PMID 26135691